CLINICAL TRIAL: NCT07320170
Title: Evaluation of the Effects of Platelet-rich Plasma and Concentrated Growth Factor on Postoperative Pain, Swelling, and Alveolar Osteitis After Mandibular Third Molar Surgery: a Randomized Controlled Clinical Trial
Brief Title: Comparative Effects of CGF and PRP in Impacted Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Emin Valiyev, Principal Investigator, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/52
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Impacted Third Molar
Keywords: Third Molar Surgery; PRP; CGF

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Standard surgical extraction was performed without the application of any additional biomaterials.
- CGF Group (Experimental): Standard surgical extraction followed by the placement of a Concentrated Growth Factor (CGF) clot into the extraction socket.
  Interventions: Biological: Concentrated Growth Factor (CGF)
- PRP Group (Experimental): Standard surgical extraction followed by submucosal injection of Platelet-Rich Plasma (PRP).
  Interventions: Biological: Platelet-Rich Plasma (PRP)

INTERVENTIONS:
Biological: Concentrated Growth Factor (CGF) — Standard surgical extraction followed by the placement of a Concentrated Growth Factor (CGF) clot into the extraction socket immediately after tooth removal.
  Arms: CGF Group
Biological: Platelet-Rich Plasma (PRP) — Standard surgical extraction followed by submucosal injection of Platelet-Rich Plasma (PRP) around the extraction site.
  Arms: PRP Group

SUMMARY:
This study evaluates the effects of two different blood products obtained from the patient's own blood (Concentrated Growth Factor [CGF] and Platelet-Rich Plasma [PRP]) on healing after wisdom tooth extraction. The aim is to determine whether applying these materials to the extraction area reduces postoperative pain, facial swelling, and the risk of dry socket compared to standard healing.

DETAILED DESCRIPTION:
This prospective, randomized, controlled clinical trial compares the efficacy of autologous platelet concentrates in reducing postoperative sequelae following the surgical extraction of impacted mandibular third molars.

A total of 42 patients were randomly assigned to one of three groups:

Control Group: Standard surgical extraction without additional biomaterials.

CGF Group: Standard extraction followed by the placement of a CGF clot into the extraction socket.

PRP Group: Standard extraction followed by submucosal injection of PRP.

The primary outcome measured is postoperative pain (Visual Analog Scale) on postoperative days 1, 3, and 7. The secondary outcomes include facial swelling (linear measurements) on postoperative days 1, 3, and 7, and the incidence of alveolar osteitis (dry socket).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 50 years.
* Systemically healthy individuals classified as American Society of Anesthesiologists (ASA) Class I or Class II.
* Presence of impacted mandibular third molars (teeth 38 and 48 according to Fédération Dentaire Internationale (FDI) notation).
* Mesioangular impaction with bone retention according to Winter's classification.
* Class II relationship to the ramus according to the Pell and Gregory classification.
* Level B or Level C depth of impaction according to the Pell and Gregory classification.

Exclusion Criteria:

* Patients younger than 18 years.
* Habitual smoking or alcohol consumption.
* Presence of coagulation (bleeding) disorders.
* Systemic diseases affecting wound healing or use of medications that compromise healing.
* Pregnancy or lactation.
* Presence of active pericoronitis associated with the tooth.
* Presence of pathological lesions (cysts or tumors) associated with the impacted tooth.
* Uncontrolled periodontal disease in the oral cavity.
* Known allergy to any medications used in the study protocol.
* Inability to comply with follow-up visits.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperative days 1, 3, and 7.
  Assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Facial Swelling | Preoperative and Postoperative days 1, 3, and 7.
  Measured using linear distances between specific facial landmarks (tragus to mouth commissure, tragus to pogonion, lateral canthus to mandibular angulus) to evaluate edema.
Incidence of Alveolar Osteitis | Postoperative days 1, 3, and 7
  Evaluated based on clinical signs such as loss of blood clot, intense throbbing pain, and halitosis (dry socket).

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University, Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.